CLINICAL TRIAL: NCT04100694
Title: Treatment Plan of the HER2/HER3 Bispecific Antibody, MCLA-128, for a Patient With Advanced NRG1-Fusion Positive Solid Tumor
Brief Title: Early Access Program Providing HER2/HER3 Bispecific Antibody, MCLA-128, for a Patient With Advanced NRG1-Fusion Positive Solid Tumor
Status: Approved for marketing | Type: Expanded Access
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: MCLA-128-CL99; MCLA-128-CL98
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: NRG1 Fusion; Pancreatic Cancer; Non Small Cell Lung Cancer; Solid Tumor, Unspecified, Adult; Prostate Cancer; Head and Neck Cancer; Colorectal Cancer; Breast Cancer; Cholangiocarcinoma; Renal Cell Carcinoma; Unknown Primary Tumors
Keywords: Early Access; NRG1 fusion; Pancreas cancer; Non Small Cell Lung Cancer; Solid tumor; Compassionate use; Expanded access
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Head and Neck Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Cholangiocarcinoma; Carcinoma, Renal Cell; Neoplasms, Unknown Primary | interventions — zenocutuzumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: MCLA-128

SUMMARY:
Merus is providing single patient/named access to the HER2/HER3 bispecific antibody, MCLA-128, to patients with advanced NRG1-fusion positive solid tumor under this early access program who are ineligible for an ongoing MCLA-128 clinical trial or have other considerations that prevent access to MCLA-128 through an existing clinical trial. Participating sites will be added as they apply for and are approved for the EAP. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* At least one evaluable or measurable lesion according to RECIST v1.1
* Patient with advanced metastatic solid tumor with documented NRG1 fusion determined in a qualified local laboratory by molecular profiling using methods such as next generation sequencing [DNA or RNA] as routinely performed at CLIA or other similarly-certified laboratories.
* Treatment with anticancer medications or investigational drugs within the following intervals before the first administration of MCLA-128:

  1. At least 14 days for chemotherapy, targeted small molecule therapy, or radiation therapy OR
  2. At least 5 half-lives have passed since discontinuation of the systemic treatment
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Adequate organ function at the time of initiation of treatment administration
* Negative pregnancy test results in women of childbearing potential (defined as women ≤50 years of age or history of amenorrhea for ≤12 months prior to study entry)
* Ability to give written, informed consent prior to treatment, with the understanding that the consent may be withdrawn by the patient at any time without prejudice
* Not eligible or feasible to participate in a clinical trial
* Any condition that in the opinion of Merus may preclude appropriate use of the investigational medicine

Exclusion Criteria:

* Any untreated, symptomatic central nervous system (CNS) lesion
* Presence of an active and uncontrolled infection
* Leptomeningeal metastases
* Known hypersensitivity to any of the components of MCLA-128 or history of severe hypersensitivity reactions to human or humanized monoclonal antibodies, including therapeutic antibodies
* Presence of LVEF <50% on the screening echocardiogram; or history or presence of any significant cardiovascular disease, including unstable angina or myocardial infarction within 12 months prior to treatment, congestive heart failure (NYHA Class III or IV), or ventricular arrhythmia requiring medication
* Presence of any other medical or psychological condition deemed by the Physician to be likely to interfere with a patient's ability to sign informed consent, cooperate or participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult